CLINICAL TRIAL: NCT00127244
Title: Outcomes of Traditional and Medical Models of Periodontal Therapy
Brief Title: Study Comparing Two Different Methods of Treating Periodontal Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Forsyth Institute (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); Delta Dental Plan Massachusetts (Unknown); Harvard University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIDCR-13850; R01DE013850 (NIH); DE-013850
Record Dates: First submitted 2005-08-04; First posted 2005-08-05 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-11

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases | interventions — Periodontal Index

INTERVENTIONS:
Procedure: Periodontal Treatment

SUMMARY:
The purposes of this study are to:

1. compare the clinical effectiveness of a traditional and a medical model of periodontal therapy; and
2. determine the value of the two approaches to periodontal therapy.

DETAILED DESCRIPTION:
This application was developed to test the following hypothesis: A medical model of periodontal therapy, when compared to a traditional model, is as clinically effective, is more valuable, and can be realistically implemented in clinical practice. To accomplish this task a prospective, blinded, community based, cohort trial will be carried out. Two analytical techniques will be employed to compare the outcomes of periodontal therapy: clinical effectiveness and value. The two primary outcome variables for assessing clinical effectiveness will be clinician centered (attachment level) and patient centered (quality of life). The key outcome variable for value determination is cost of care. Value is then determined by dividing the outcome by the cost of care. Thus a similar outcome at reduced cost increases value. This facilitates calculating cost-effectiveness and cost-utility of care, preparing decision analysis trees, and carrying out sensitivity analysis.

There are two significant reasons for testing a medical model of care. If the hypothesis is correct:

1. this would increase access to periodontal care; and
2. it would offer a cost-effective method to treat periodontal infections that are correlated with systemic health problems.

These points argue for a direct comparison of the medical and traditional models of care.

ELIGIBILITY:
Inclusion Criteria:

* >/= 4 or more periodontally involved teeth as defined by pocket depth of >/= 6mm.
* >/= 14 teeth.
* > 18 years of age.
* Reside in the greater Boston area.

Exclusion Criteria:

* Those patients requiring prophylactic antibiotic for dental treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2000-06; Study Completion 2004-10

PRIMARY OUTCOMES:
Clinical attachment loss
Quality of life
Tooth loss
Plaque accumulation
Suppuration
Bleeding on probing

CONTACTS AND LOCATIONS:
Overall Officials: Richard Niederman, Principal Investigator — The Forsyth Institute
Locations (1):
- The Forsyth Institute, Boston, Massachusetts, United States